CLINICAL TRIAL: NCT06288724
Title: Potentially MOdifiable Factors To ImproVe Outcomes of Mechanically Ventilated Patients in ICUs in a Low-income Country: Rationale and Protocol for a Registry-embedded Prospective Observational Study
Brief Title: MOdifiable facTors to Improve VentilAtion ThErapy in ICU
Acronym: MOTIVATE-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Nat Intensive Care Surveillance - MORU (Other)
Collaborators: D'Or Institute for Research and Education (Other); University of Oxford (Other); Wellcome Trust (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Cornelius Sendagire, DR, Nat Intensive Care Surveillance - MORU
Other Study IDs: NatIntensive
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness; Invasive Mechanical Ventilation; ICU Mortality; Developing Countries; Risk Factors
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ABSTRACT Introduction: Invasively ventilated patients in low and middle-income countries (LMICs) experience significantly higher mortality compared to those in High income countries (HICs). Direct application of HIC strategies to LMICs maybe ineffective due to context-specific challenges. This study aims to leverage the Intensive Care Registry of Uganda (ICRU) to identify ICU structural and process-related modifiable factors that impact patient outcomes in a low income country.

Methods: The MOTIVATE-ICU is a prospective multicentre observational study in invasively ventilated patients. It involves a registry-embedded component examining patient- and process-related factors and a cross-sectional survey on ICU organizational structures. Inclusion criteria encompass patients aged ≥ 15 years undergoing IMV in Ugandan ICUs. Primary outcomes are ICU mortality, ICU length of stay (LOS), and duration of ventilation. Secondary outcomes include ventilator-associated complications, non-pulmonary organ support. tTracheostomy outcomes will be explored in a pre-planned substudy. Factors potentially associated with outcomes will be categorized into two groups; non-modifiable factors and potentially modifiable. Non-modifiable factors will include patient-related factors like age, comorbidities and illness severity; potentially modifiable factors include processes of care (e.g. sedation levels) and ICU organizational structure (e.g. staffing patterns). Multilevel multivariable logistic regression will be utilized to study associations, with both patient and ICU level fixed effects considered.

Ethics and Dissemination: Given its observational nature, this study seeks a waiver for patient individual informed consent. Data anonymization ensures patient privacy. Following the principles of the Declaration of Helsinki, relevant ethical approvals will be acquired. Study findings will be disseminated through conferences and peer-reviewed journals.

DETAILED DESCRIPTION:
Introduction:

In low and middle-income countries (LMICs), up to two-thirds of ICU admissions necessitate invasive mechanical ventilation (IMV), compared to half of ICU admissions globally1-3. Though IMV is a life saving organ support technique, it's also linked to complications like ventilator associated lung injury and requires complex processes of care4. Despite being younger, ventilated patients in LMICs have 2-4 times higher mortality than high-income countries (HICs)5-8. Patients with acute respiratory distress syndrome (ARDS) in LMICs face an even greater risk, 70% higher than in HICs9.

While HICs have ample data on modifiable factors and improvement strategies that curtail ICU complications, LMICs may face preventable complications associated with IMV1,10-13. Complications like ventilator-induced lung injury and related pneumonia lead not only to excess deaths but also longer ICU stays and escalating costs14. Unfortunately, data on determinants of poor outcome among ventilated patients in LMICs remains scarce 12,15-17. Directly applying HIC evidence based management strategies to LMICs isn't always effective, as seen in several African trials 18,19. LMICs grapple with challenges like understaffing, limited training, insufficient infrastructure, and different patient characteristics and comorbidities, all potentially compromising the quality of ICU care15,16,20,21.

Recently, the use of critical care registries for data collection, including patient care, indicators, and outcomes, has expanded in both HICs and LMICs22-24. This streamlines research and offers cost benefits. Uganda has launched the Intensive Care Registry of Uganda (ICRU) for quality improvement and research infrastructure. This registry-embedded study aims to identify modifiable factors impacting outcomes for mechanically ventilated patients in LMICs leveraging ICRU's data pipeline. We hypothesize that specific patient-level and organizational factors can be identified that contribute to the ICU mortality of ventilated patients in Uganda.

Methods and Analysis:

Study design:

The 'Potentially MOdifiable factors To ImproVe outcomes of mechanically Ventilated patients in ICUs in a Low-income Country' (MOTIVATE-ICU) study is a prospective multicentre registry-embedded observational study with two main components. The first will be a prospective observational multicenter registry-embedded study aimed at assessing patient-related and process-related factors. The second component will be a cross-sectional survey to assess the organizational structure of the ICUs included. This study protocol was registered at Clinicaltrials.gov (registration number: NCTXXXXXXX). The results of the study will be reported according to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement25.

Study setting:

ICUs will be defined as geographically designated area/unit within a hospital that routinely provides invasive mechanical ventilation therapy with continuous vital sign monitoring [electrocardiographic (ECG) monitoring, heart/pulse rate, non-invasive blood pressure (NIBP), peripheral oxygen saturation (SpO2)] and designated nursing care for each bed in the unit i.e at least three patients per week for at least 24 hours. A descriptive study conducted in Uganda assessing the ICU capacity before the Corona virus induced disease 2019 (COVID-19) revealed that at the time, there were 14 ICUs with 12 being functional20. However, post-COVID-19, anecdotal evidence shows nearly a doubling of the ICU capacity with nearly 25 functional ICUs to-date. All ICUs currently functional in Uganda will be eligible to participate (eTable 1).

Participants:

Patients aged ≥ 15 years admitted to study ICUs during the study period and receiving invasive mechanical ventilation will be eligible for recruitment. Exclusion criteria include successful extubations within 24 hours of intubation, admissions for end-of-life care and/or ICU palliative support as well as patients transferred from ICUs not participating in the study 24 hours after initiation of MV.

Outcomes:

Primary outcomes The primary outcomes will be ICU mortality, ICU length of stay (LOS) and duration of mechanical ventilation. Outcome definitions are detailed in Table 1.

Secondary outcomes These will include duration of non-pulmonary organ support, ICU-free days, ventilator-free days at day 28, ventilator-associated pneumonia (VAP), tracheobronchitis, non-infectious pulmonary complication (clinician suspicion or radiological diagnosis of pleural effusion, atelectasis or pneumothorax), readmission, unplanned extubations. Tracheostomy related outcomes will be explored as part of a preplanned substudy, including tracheostomy timing, decannulation rate, decannulation failure and complications such as stoma infection, major bleeding, tube dislodgement and malfunction.

Associated factors (Table 2):

Factors potentially associated with outcomes among mechanically ventilated patients will be analyzed as 'non-modifiable' factors and 'potentially modifiable' factors. Non-modifiable factors include patient-related factors such as age, illness severity at initiation of mechanical ventilation, comorbidities, medical vs surgical admission, and indication for IMV (Table 2). Potentially modifiable factors will subcategorized into care process-related factors such as Richmond Agitation Sedation Scale (RASS) targets, initial ventilator settings on day 0, use of daily spontaneous awakening and spontaneous breathing trials, use of stress ulcer and deep vein thrombosis (DVT) prophylaxis. The second subcategory will be ICU organizational structure such ICU staffing, staff-patient ratios, empowerment of non-physician staff, multidisciplinary team rounds and use of protocols and checklists (Details on associated factors in supplementary material Table 2).

Data collection:

The following procedures will be performed to ensure the quality of the data collection Patient-level data will be entered directly via laptop or tablet through the cloud-based ICU registry platform (PROTECT cloud-based platform) of the ICRU currently in use (Figure 1).

Patient level variables of interest including age, sex, diagnostic categories, functional capacity before hospital admission (Clinical Frailty Score), the Charlson Comorbidity Index, the use of IMV on Day 1, modified Sequential Organ Function Assessment (mSOFA) and Tropical Intensive Care Score (e-TropICS) will be scored. ICU level variables of interest included ICU type (medical-surgical vs. specialty), presence of training programs in critical care, ICU admission volumes in the preceding year, staffing patterns, organizational and process characteristics; a full list of potential covariates is detailed in Table 2.

We shall extract prospectively collected data from the ICRU platform, which has both core data variables collected at admission and daily variables collected during the ICU stay.

A complete list of variables is detailed in Supplementary materials. The platform uses a common data model and provides real-time data on casemix, management features and outcomes. MOTIVATE-ICU study variables were incorporated into the PROTECT platform in order to design a registry embedded study (Figure 1). The following site-level procedures will be followed:

To ensure standardization of the study procedures, each site shall have a site lead and dedicated data entrant(s) responsible for data collection during use of the ICU registry platform. Prior to the beginning of recruitment, each site lead and data entrant(s) will receive training.

Each site will have a site lead responsible for weekly validation of patient episodes in terms of completion and data quality.

Each site will have IT support as well as participate in monthly meetings as a means of dispelling doubts and solving potential challenges related to data entry.

For each site, data on hospital and ICU organizational and care process characteristics will be collected through an interviewer-administered questionnaire from the ICU director and/or the in-charge nurse.

Follow-up:

Given the potential burden of data collection involved, the patient recruitment period in each participating ICU will be a minimum of three months up to a maximum of 6 months, with a 28-day maximum follow-up period for each patient recruited. The follow up period for individual patients will end at ICU discharge.

Procedures to ensure data quality

Sample size:

We aim to include all consecutive patients admitted to participating ICUs in order to reduce potential selection bias and minimise temporal variation of care processes. Based on aggregated data (published and unpublished) from LMICs including Uganda's ICU cohorts2,10,12,26-31 the lowest measured mortality among patients receiving invasive mechanical ventilation was approximately 40%. A total of 250 events (deaths) would allow us to evaluate at least 25 associated variables in multivariable models. We will therefore enroll at least 625 patients receiving invasive mechanical ventilation that fulfill the eligibility criteria.

Handling of missing data:

During the study period, all data pertinent to the study objectives will be mandated for all study ICUs. The study platform will flag missing data to the data collector in case of incompleteness. Each site lead will ensure validation of patients entered and completeness of the data weekly to ensure no missing data. This is being a prospective registry-embedded study, we expect a low percentage of missing data pertinent to the primary objectives of the study.

Statistical analysis:

We will describe ICU and patient characteristics using standard descriptive statistics and reported continuous variables as mean ± standard deviation or median (25%-75% interquartile range, IQR), as appropriate. We will test the univariate association between eligible variables and outcomes using analysis of variance, Kruskal-Wallis, Student t test, Mann-Whitney test, chi-square test, and Fisher exact test, as appropriate.

Using multilevel multivariable logistic regression models, we shall investigate the association between organizational factors and the primary outcome adjusting for patients' characteristics. A two-level model will be fit with patient-level fixed effects at the first level and ICU-level fixed effects at the second level, as well as an ICU-specific random effect. We will pre-specify several models to represent the patients and the unit organization dimensions. We shall then insert variables into the models if they are associated with outcome with a P value of <0.20 on univariate analysis. We shall not consider variables used for e-TropICS score computation. We shall apply several variables into the final model regardless of their statistical significance due to their clinical significance, including the presence of 24/7 intensivist, regular multidisciplinary rounds and nurse/bed ratios in the final model. In addition, we shall perform subgroup analyses stratifying patients according to the type of admission (medical vs. surgical) and the e-TropICS tertiles. We shall use the Akaike information criterion, the likelihood ratios and the model residuals to choose among the alternative models. Two-tailed P-values <0.05 were considered statistically significant. All statistical analyses will be conducted in R (http://www.r-project.org) and SPSS 21 (IBM Corp., Armonk, NY). A detailed statistical analysis plan will be made available online before completion of the study and locking of the database.

Ethics and dissemination:

Ethical approval and consent to participate This study will be conducted according to the principles of the Declaration of Helsinki (revision Fortaleza, Brazil, October 2013). Approval to carry out this study will be sought from the relevant ethical review and scientific review committees and from hospital administrations.

We shall obtain deferred consent within 72 hours of recruitment into the study from the legal representative since most ICU admissions are emergency admissions and informed consent during the initial 48 hours of admission may not be possible. In addition, without exception, patients admitted to ICU for ventilator support are unable to give informed consent. Persons who may take the role of legal representative in accordance with the Medical Treatment Agreement Act (WGBO) are: a predefined representative, husband or wife, registered partner or other life partner, a parent or child, brother or sister, and incidentally a curator appointed by a judge. For patients with no legal representative and are unable to give informed consent during in-hospital stay, we shall obtain a waiver of consent. The experience of ICU patients enrolled under deferred consent is mainly positive, as shown in the NICE-SUGAR trial, in which participants were included using deferred consent32. A majority of the patients were happy with the decision made by the representative (93%) and would have granted consent if asked (96%)33.

Oral consent from each of the ICU directors and/or in-charge nurse will be sought to conduct the interviewer-administered survey.

Dissemination:

The study results will be submitted for publication regardless of the results after completion and analysis. We shall make the study findings widely available including dissemination through conferences and peer-reviewed journals.

Data sharing:

The authors encourage interested parties to contact the corresponding author with data sharing requests, including for access to additional unpublished data. ICRU is part of a larger network which has appointed a Data Access Committee (DAC). Curated data may be shared with third parties for research purposes following written approval from the DAC.

Discussion and study status:

The MOTIVATE-ICU registry-embedded study aims to identify potentially modifiable factors associated with outcomes among invasively ventilated patients in a low income country.

According to the Donabedian model improving the quality of healthcare and improving outcomes of interest, rests on three components; the structure, care processes and outcomes.34 Various studies from HICs on ICU organization structure, care-bundles and protocols have shown significant impact in reduction of mortality, duration of ventilation and ICU length of stay; albeit with some inconsistencies in some aspects.6,11,35-37 Based on what we currently know from the ORCHESTRA study done in Brazil, an upper middle income country (UMIC), organizational factors including protocol implementation are the key targets to improve ICU outcomes and efficiency38,39. There has been considerable data describing the physical structural set-up and staffing of ICUs in LMICs20,26,40,41, but limited data is available on organizational features and care-processes, and their impact on outcomes in lower income settings like Uganda.

Direct implementation of evidence-based care processes from higher income settings may not necessarily yield similar results when implemented in resource-poor settings. For example, two African studies that implemented fluid therapy as per protocols used in HICs revealed more harm than benefit in both critically ill adults and paediatric populations18,19. For other processes, implementation in LMICs has improved consistently but outcomes remain lagging when compared to HICs, probably affected by a multitude of factors. For instance, use of protective mechanical ventilation in patients without ARDS was shown to be comparable between MICs and HICS during first days of ventilation, but with a large difference in ICU mortality14. The same was seen for ventilation in ARDS patients, albeit with a small difference in protective ventilation implementation1,6.

One of the key potential interventions likely to show impact in low-resource settings compared to HICs is tracheostomy placement and timing. Tracheostomy timing, while improving ICU length of stay and duration of mechanical ventilation has not had an impact on mortality in HICs42-44, but may have a significant impact in a setting with limited resources. A preplanned substudy of MOTIVATE-ICU will explore timing, complications and outcomes in patients undergoing tracheostomy in a low income country like Uganda, complementing data from LMICs from other African countries45,46.

The strengths of the current study are its prospective design, registry-embedded nature, and multicenter inclusion. There are several potential limitations of this study. For example, while efforts are made to ensure data quality and reduce missing data, the reliance on electronic data collection and the prospective nature of the study may still encounter challenges with data completeness and accuracy across multiple centers. The study's findings, especially those related to organizational structure and process-related factors, may be specific to the context of low-income countries and thus may not be generalizable to settings with different healthcare systems, resources, and ICU capabilities. The cross-sectional survey assessing the organizational structure of ICUs, rely on self-reported data, which can introduce biases and inaccuracies.

Acknowledgements:

We thank all the site leads and data entrants of each site at each of the participating hospitals as well as Critical Care Asia Africa network for the support and involvement in the success of this study.

Funding:

The study will be supported by the Wellcome award, Collaboration for Research, Implementation and Training in Critical Care in Asia and Africa (Grant number: 224048/Z/21/Z).

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilatory support initiated anywhere within the study hospital i.e., emergency room, normal ward or in the operating room, or in the ICU at any time during admission.

Exclusion Criteria:

* Successful extubations within two calendar days of intubation
* Admissions for end-of-life care and/or ICU palliative support
* Patients transferred from ICUs not participating in the study 24 hours after initiation of MV.
* Refusal or Withdrawal of consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥15 years receiving invasive mechanical ventilation within the ICU
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 28 days
  Death at ICU discharge, or at 28 days after ICU admission, whichever occurs first.
ICU Length of Stay | 28 days
  Number of days patients spend in the ICU. Measured per episode of ICU care. Calculated using the interval (measured in hours) between the date and time of ICU admission and the date and time of ICU discharge. Rounded to the nearest 1 decimal place.
Duration of mechanical ventilation | 28 days
  The time between endotracheal intubation and successful extubation (in case of intermittent mechanical ventilation via a tracheostomy, every day a patient needs ventilation counts as one extra day, irrespective of the duration of ventilation on that specific day). In case of non-invasive ventilation, the duration will be assessed separated from the assessment of invasive ventilation.

SECONDARY OUTCOMES:
Duration of non-pulmonary organ support | 28 days
  Time between initiation of vasopressor/inotropic support or renal replacement therapy to the time of discontinuation for at least 24 hours. Individual components of the composite outcome will be reported.
ICU-Free days | 28 days
  Number of in-hospital days from ICU discharge to 28 days. If the patient dies after ICU discharge and before 28 days this will count as 0
Ventilator-free days | 28 days
  The number of ventilator-free days at 28 days (VFD-28) will be determined by subtracting the total duration of mechanical ventilation from 30 days. If a patient passed away before reaching the 28-day mark, their VFD-28 will be recorded as having zero VFD-28
Ventilator-associated Pneumonia | 28 days
  Presence of fever OR Altered leukocyte count PLUS New onset of purulent endotracheal secretions OR change in sputum WITH new and progressive or persistent infiltrate or consolidation or cavitation48 For those without radiological diagnosis, we shall consider clinically suspected VAP.
Tracheobronchitis | 28 days
  Presence of fever OR altered leukocyte count (<4 or >12 x 103) PLUS New onset of purulent endotracheal secretions OR change in sputum
Non-infectious Pulmonary complication | 28 days
  Clinician suspicion or radiological diagnosis of pleural effusion, atelectasis or pneumothorax
Readmission | 28 days
  Unplanned ICU admission within 48 hours after ICU discharge
Unplanned extubations | 28 days
  Inadvertent/accidental extubations requiring reintubation
Tracheostomy related outcomes | 28 days
  The following outcomes will be included:
  Timing of tracheostomy in terms of number of days after intubation; decannulation rate, i.e. the proportion of patients undergoing successful decannulation during ICU stay decannulation failure (defined as the need to recannulate for any reason between decannulation and hospital discharge); Tracheostomy-related complications: stoma infection, major bleeding, tube dislodgement, and malfunction defined as air leaks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laffey JG, Bellani G, Pham T, Fan E, Madotto F, Bajwa EK, Brochard L, Clarkson K, Esteban A, Gattinoni L, van Haren F, Heunks LM, Kurahashi K, Laake JH, Larsson A, McAuley DF, McNamee L, Nin N, Qiu H, Ranieri M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators and the ESICM Trials Group. Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study. Intensive Care Med. 2016 Dec;42(12):1865-1876. doi: 10.1007/s00134-016-4571-5. Epub 2016 Oct 18. PMID 27757516
- [Background] Prin M, Itaye T, Clark S, Fernando RJ, Namboya F, Pollach G, Mkandawire N, Sobol J. Critical Care in a Tertiary Hospital in Malawi. World J Surg. 2016 Nov;40(11):2635-2642. doi: 10.1007/s00268-016-3578-y. PMID 27230398
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] Goligher EC, Ferguson ND, Brochard LJ. Clinical challenges in mechanical ventilation. Lancet. 2016 Apr 30;387(10030):1856-66. doi: 10.1016/S0140-6736(16)30176-3. Epub 2016 Apr 28. PMID 27203509
- [Background] Inglis R, Ayebale E, Schultz MJ. Optimizing respiratory management in resource-limited settings. Curr Opin Crit Care. 2019 Feb;25(1):45-53. doi: 10.1097/MCC.0000000000000568. PMID 30531535
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Neto AS, Barbas CSV, Simonis FD, Artigas-Raventos A, Canet J, Determann RM, Anstey J, Hedenstierna G, Hemmes SNT, Hermans G, Hiesmayr M, Hollmann MW, Jaber S, Martin-Loeches I, Mills GH, Pearse RM, Putensen C, Schmid W, Severgnini P, Smith R, Treschan TA, Tschernko EM, Melo MFV, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ; PRoVENT; PROVE Network investigators. Epidemiological characteristics, practice of ventilation, and clinical outcome in patients at risk of acute respiratory distress syndrome in intensive care units from 16 countries (PRoVENT): an international, multicentre, prospective study. Lancet Respir Med. 2016 Nov;4(11):882-893. doi: 10.1016/S2213-2600(16)30305-8. Epub 2016 Oct 4. PMID 27717861
- [Background] Khatib KI, Dixit SB, Joshi MM. Factors determining outcomes in adult patient undergoing mechanical ventilation: A "real-world" retrospective study in an Indian Intensive Care Unit. Int J Crit Illn Inj Sci. 2018 Jan-Mar;8(1):9-16. doi: 10.4103/IJCIIS.IJCIIS_41_17. PMID 29619334
- [Background] Laffey JG, Madotto F, Bellani G, Pham T, Fan E, Brochard L, Amin P, Arabi Y, Bajwa EK, Bruhn A, Cerny V, Clarkson K, Heunks L, Kurahashi K, Laake JH, Lorente JA, McNamee L, Nin N, Palo JE, Piquilloud L, Qiu H, Jimenez JIS, Esteban A, McAuley DF, van Haren F, Ranieri M, Rubenfeld G, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Geo-economic variations in epidemiology, patterns of care, and outcomes in patients with acute respiratory distress syndrome: insights from the LUNG SAFE prospective cohort study. Lancet Respir Med. 2017 Aug;5(8):627-638. doi: 10.1016/S2213-2600(17)30213-8. Epub 2017 Jun 15. PMID 28624388
- [Background] African COVID-19 Critical Care Outcomes Study (ACCCOS) Investigators. Patient care and clinical outcomes for patients with COVID-19 infection admitted to African high-care or intensive care units (ACCCOS): a multicentre, prospective, observational cohort study. Lancet. 2021 May 22;397(10288):1885-1894. doi: 10.1016/S0140-6736(21)00441-4. PMID 34022988
- [Background] Simonis FD, Barbas CSV, Artigas-Raventos A, Canet J, Determann RM, Anstey J, Hedenstierna G, Hemmes SNT, Hermans G, Hiesmayr M, Hollmann MW, Jaber S, Martin-Loeches I, Mills GH, Pearse RM, Putensen C, Schmid W, Severgnini P, Smith R, Treschan TA, Tschernko EM, Vidal Melo MF, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ, Neto AS; PRoVENT investigators; PROVE Network investigators. Potentially modifiable respiratory variables contributing to outcome in ICU patients without ARDS: a secondary analysis of PRoVENT. Ann Intensive Care. 2018 Mar 21;8(1):39. doi: 10.1186/s13613-018-0385-7. PMID 29564726
- [Background] Karthikeyan B, Kadhiravan T, Deepanjali S, Swaminathan RP. Case-Mix, Care Processes, and Outcomes in Medically-Ill Patients Receiving Mechanical Ventilation in a Low-Resource Setting from Southern India: A Prospective Clinical Case Series. PLoS One. 2015 Aug 11;10(8):e0135336. doi: 10.1371/journal.pone.0135336. eCollection 2015. PMID 26262995
- [Background] Dijkema LM, Dieperink W, van Meurs M, Zijlstra JG. Preventable mortality evaluation in the ICU. Crit Care. 2012 Dec 12;16(2):309. doi: 10.1186/cc11212. PMID 22546292
- [Background] Pisani L, Algera AG, Neto AS, Azevedo L, Pham T, Paulus F, de Abreu MG, Pelosi P, Dondorp AM, Bellani G, Laffey JG, Schultz MJ; ERICC study investigators; LUNG SAFE study investigators; PRoVENT study investigators; PRoVENT-iMiC study investigators. Geoeconomic variations in epidemiology, ventilation management, and outcomes in invasively ventilated intensive care unit patients without acute respiratory distress syndrome: a pooled analysis of four observational studies. Lancet Glob Health. 2022 Feb;10(2):e227-e235. doi: 10.1016/S2214-109X(21)00485-X. Epub 2021 Dec 13. PMID 34914899
- [Background] Vukoja M, Riviello E, Gavrilovic S, Adhikari NK, Kashyap R, Bhagwanjee S, Gajic O, Kilickaya O; CERTAIN Investigators. A survey on critical care resources and practices in low- and middle-income countries. Glob Heart. 2014 Sep;9(3):337-42.e1-5. doi: 10.1016/j.gheart.2014.08.002. Epub 2014 Oct 31. PMID 25667185
- [Background] Murthy S, Leligdowicz A, Adhikari NK. Intensive care unit capacity in low-income countries: a systematic review. PLoS One. 2015 Jan 24;10(1):e0116949. doi: 10.1371/journal.pone.0116949. eCollection 2015. PMID 25617837
- [Background] Mendsaikhan N, Begzjav T, Lundeg G, Dunser MW. Potentially Preventable Deaths by Intensive Care Medicine in Mongolian Hospitals. Crit Care Res Pract. 2016;2016:8624035. doi: 10.1155/2016/8624035. Epub 2016 Oct 4. PMID 27795857
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] Andrews B, Semler MW, Muchemwa L, Kelly P, Lakhi S, Heimburger DC, Mabula C, Bwalya M, Bernard GR. Effect of an Early Resuscitation Protocol on In-hospital Mortality Among Adults With Sepsis and Hypotension: A Randomized Clinical Trial. JAMA. 2017 Oct 3;318(13):1233-1240. doi: 10.1001/jama.2017.10913. PMID 28973227
- [Background] Atumanya P, Sendagire C, Wabule A, Mukisa J, Ssemogerere L, Kwizera A, Agaba PK. Assessment of the current capacity of intensive care units in Uganda; A descriptive study. J Crit Care. 2020 Feb;55:95-99. doi: 10.1016/j.jcrc.2019.10.019. Epub 2019 Nov 4. PMID 31715537
- [Background] GBD 2015 Healthcare Access and Quality Collaborators. Electronic address: cjlm@uw.edu; GBD 2015 Healthcare Access and Quality Collaborators. Healthcare Access and Quality Index based on mortality from causes amenable to personal health care in 195 countries and territories, 1990-2015: a novel analysis from the Global Burden of Disease Study 2015. Lancet. 2017 Jul 15;390(10091):231-266. doi: 10.1016/S0140-6736(17)30818-8. Epub 2017 May 18. PMID 28528753
- [Background] Aryal D, Beane A, Dondorp AM, Green C, Haniffa R, Hashmi M, Jayakumar D, Marshall JC, McArthur CJ, Murthy S, Webb SA, Acharya SP, Ishani PGP, Jawad I, Khanal S, Koirala K, Luitel S, Pabasara U, Paneru HR, Kumar A, Patel SS, Ramakrishnan N, Salahuddin N, Shaikh M, Tolppa T, Udayanga I, Umrani Z. Operationalisation of the Randomized Embedded Multifactorial Adaptive Platform for COVID-19 trials in a low and lower-middle income critical care learning health system. Wellcome Open Res. 2021 Jan 28;6:14. doi: 10.12688/wellcomeopenres.16486.1. eCollection 2021. PMID 33604455
- [Background] Vijayaraghavan BKT, Venkatraman R, Ramakrishnan N. Critical Care Registries: The Next Big Stride? Indian J Crit Care Med. 2019 Aug;23(8):387. doi: 10.5005/jp-journals-10071-23227. PMID 31485112
- [Background] Pisani L, Waweru-Siika W, Sendagire C, Beane A, Haniffa R. Critically ill COVID-19 patients in Africa: it is time for quality registry data. Lancet. 2021 Aug 7;398(10299):485-486. doi: 10.1016/S0140-6736(21)01549-X. No abstract available. PMID 34364515
- [Background] Cuschieri S. The STROBE guidelines. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S31-S34. doi: 10.4103/sja.SJA_543_18. PMID 30930717
- [Background] Kwizera A, Dunser M, Nakibuuka J. National intensive care unit bed capacity and ICU patient characteristics in a low income country. BMC Res Notes. 2012 Sep 1;5:475. doi: 10.1186/1756-0500-5-475. PMID 22937769
- [Background] Riviello ED, Letchford S, Achieng L, Newton MW. Critical care in resource-poor settings: lessons learned and future directions. Crit Care Med. 2011 Apr;39(4):860-7. doi: 10.1097/CCM.0b013e318206d6d5. PMID 21297458
- [Background] Sendagire C, Lipnick MS, Kizito S, Kruisselbrink R, Obua D, Ejoku J, Ssemogerere L, Nakibuuka J, Kwizera A. Feasibility of the modified sequential organ function assessment score in a resource-constrained setting: a prospective observational study. BMC Anesthesiol. 2017 Jan 26;17(1):12. doi: 10.1186/s12871-017-0304-8. PMID 28122489
- [Background] Ttendo SS, Was A, Preston MA, Munyarugero E, Kerry VB, Firth PG. Retrospective Descriptive Study of an Intensive Care Unit at a Ugandan Regional Referral Hospital. World J Surg. 2016 Dec;40(12):2847-2856. doi: 10.1007/s00268-016-3644-5. PMID 27506722
- [Background] Parker RK, Mwachiro EB, Mwachiro MM, Pletcher J, Parker AS, Many HR. Mortality Prediction in Rural Kenya: A Cohort Study of Mechanical Ventilation in Critically Ill Patients. Crit Care Explor. 2019 Dec 10;1(12):e0067. doi: 10.1097/CCE.0000000000000067. eCollection 2019 Dec. PMID 32166248
- [Background] Towey RM, Ojara S. Intensive care in the developing world. Anaesthesia. 2007 Dec;62 Suppl 1:32-7. doi: 10.1111/j.1365-2044.2007.05295.x. PMID 17937711
- [Background] Arabi YM, Dabbagh OC, Tamim HM, Al-Shimemeri AA, Memish ZA, Haddad SH, Syed SJ, Giridhar HR, Rishu AH, Al-Daker MO, Kahoul SH, Britts RJ, Sakkijha MH. Intensive versus conventional insulin therapy: a randomized controlled trial in medical and surgical critically ill patients. Crit Care Med. 2008 Dec;36(12):3190-7. doi: 10.1097/CCM.0b013e31818f21aa. PMID 18936702
- [Background] Potter JE, McKinley S, Delaney A. Research participants' opinions of delayed consent for a randomised controlled trial of glucose control in intensive care. Intensive Care Med. 2013 Mar;39(3):472-80. doi: 10.1007/s00134-012-2732-8. Epub 2012 Oct 25. PMID 23096429
- [Background] Donabedian A. Evaluating the quality of medical care. 1966. Milbank Q. 2005;83(4):691-729. doi: 10.1111/j.1468-0009.2005.00397.x. No abstract available. PMID 16279964
- [Background] Barr J, Ghaferi AA, Costa DK, Hedlin HK, Ding VY, Ross C, Pun BT, Watson SR, Asch SM. Organizational Characteristics Associated With ICU Liberation (ABCDEF) Bundle Implementation by Adult ICUs in Michigan. Crit Care Explor. 2020 Aug 19;2(8):e0169. doi: 10.1097/CCE.0000000000000169. eCollection 2020 Aug. PMID 32885171
- [Background] Pun BT, Balas MC, Barnes-Daly MA, Thompson JL, Aldrich JM, Barr J, Byrum D, Carson SS, Devlin JW, Engel HJ, Esbrook CL, Hargett KD, Harmon L, Hielsberg C, Jackson JC, Kelly TL, Kumar V, Millner L, Morse A, Perme CS, Posa PJ, Puntillo KA, Schweickert WD, Stollings JL, Tan A, D'Agostino McGowan L, Ely EW. Caring for Critically Ill Patients with the ABCDEF Bundle: Results of the ICU Liberation Collaborative in Over 15,000 Adults. Crit Care Med. 2019 Jan;47(1):3-14. doi: 10.1097/CCM.0000000000003482. PMID 30339549
- [Background] Kerlin MP, Adhikari NK, Rose L, Wilcox ME, Bellamy CJ, Costa DK, Gershengorn HB, Halpern SD, Kahn JM, Lane-Fall MB, Wallace DJ, Weiss CH, Wunsch H, Cooke CR; ATS Ad Hoc Committee on ICU Organization. An Official American Thoracic Society Systematic Review: The Effect of Nighttime Intensivist Staffing on Mortality and Length of Stay among Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Feb 1;195(3):383-393. doi: 10.1164/rccm.201611-2250ST. PMID 28145766
- [Background] Soares M, Bozza FA, Angus DC, Japiassu AM, Viana WN, Costa R, Brauer L, Mazza BF, Correa TD, Nunes AL, Lisboa T, Colombari F, Maciel AT, Azevedo LC, Damasceno M, Fernandes HS, Cavalcanti AB, do Brasil PE, Kahn JM, Salluh JI. Organizational characteristics, outcomes, and resource use in 78 Brazilian intensive care units: the ORCHESTRA study. Intensive Care Med. 2015 Dec;41(12):2149-60. doi: 10.1007/s00134-015-4076-7. PMID 26499477
- [Background] Zampieri FG, Salluh JIF, Azevedo LCP, Kahn JM, Damiani LP, Borges LP, Viana WN, Costa R, Correa TD, Araya DES, Maia MO, Ferez MA, Carvalho AGR, Knibel MF, Melo UO, Santino MS, Lisboa T, Caser EB, Besen BAMP, Bozza FA, Angus DC, Soares M; ORCHESTRA Study Investigators. ICU staffing feature phenotypes and their relationship with patients' outcomes: an unsupervised machine learning analysis. Intensive Care Med. 2019 Nov;45(11):1599-1607. doi: 10.1007/s00134-019-05790-z. Epub 2019 Oct 8. PMID 31595349
- [Background] Haniffa R, De Silva AP, Iddagoda S, Batawalage H, De Silva ST, Mahipala PG, Dondorp A, de Keizer N, Jayasinghe S. A cross-sectional survey of critical care services in Sri Lanka: a lower middle-income country. J Crit Care. 2014 Oct;29(5):764-8. doi: 10.1016/j.jcrc.2014.04.021. Epub 2014 May 9. PMID 24929445
- [Background] Phua J, Faruq MO, Kulkarni AP, Redjeki IS, Detleuxay K, Mendsaikhan N, Sann KK, Shrestha BR, Hashmi M, Palo JEM, Haniffa R, Wang C, Hashemian SMR, Konkayev A, Mat Nor MB, Patjanasoontorn B, Nafees KMK, Ling L, Nishimura M, Al Bahrani MJ, Arabi YM, Lim CM, Fang WF; Asian Analysis of Bed Capacity in Critical Care (ABC) Study Investigators, and the Asian Critical Care Clinical Trials Group. Critical Care Bed Capacity in Asian Countries and Regions. Crit Care Med. 2020 May;48(5):654-662. doi: 10.1097/CCM.0000000000004222. PMID 31923030
- [Background] Chorath K, Hoang A, Rajasekaran K, Moreira A. Association of Early vs Late Tracheostomy Placement With Pneumonia and Ventilator Days in Critically Ill Patients: A Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2021 May 1;147(5):450-459. doi: 10.1001/jamaoto.2021.0025. PMID 33704354
- [Background] Alali AS, Scales DC, Fowler RA, Mainprize TG, Ray JG, Kiss A, de Mestral C, Nathens AB. Tracheostomy timing in traumatic brain injury: a propensity-matched cohort study. J Trauma Acute Care Surg. 2014 Jan;76(1):70-6; discussion 76-8. doi: 10.1097/TA.0b013e3182a8fd6a. PMID 24368359
- [Background] Queen Elizabeth Hospital Birmingham COVID-19 airway team. Safety and 30-day outcomes of tracheostomy for COVID-19: a prospective observational cohort study. Br J Anaesth. 2020 Dec;125(6):872-879. doi: 10.1016/j.bja.2020.08.023. Epub 2020 Aug 28. PMID 32988602
- [Background] Prin M, Kaizer A, Cardenas J, Mtalimanja O, Kadyaudzu C, Charles A, Ginde A. Tracheostomy Practices for Mechanically Ventilated Patients in Malawi. World J Surg. 2021 Sep;45(9):2638-2642. doi: 10.1007/s00268-021-06176-3. Epub 2021 Jun 2. PMID 34080049
- [Background] Mulima G, Lie SA, Charles A, Hanif AB, Varela CG, Banza LN, Young S. Tracheostomy without mechanical ventilation in patients with traumatic brain injury at a tertiary referral hospital in Malawi: a cross sectional study. Malawi Med J. 2022 Sep;34(3):152-156. doi: 10.4314/mmj.v34i3.2. PMID 36406102
- [Background] Renard Triche L, Futier E, De Carvalho M, Pinol-Domenech N, Bodet-Contentin L, Jabaudon M, Pereira B. Sample size estimation in clinical trials using ventilator-free days as the primary outcome: a systematic review. Crit Care. 2023 Aug 1;27(1):303. doi: 10.1186/s13054-023-04562-y. PMID 37528425
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Weled BJ, Adzhigirey LA, Hodgman TM, Brilli RJ, Spevetz A, Kline AM, Montgomery VL, Puri N, Tisherman SA, Vespa PM, Pronovost PJ, Rainey TG, Patterson AJ, Wheeler DS; Task Force on Models for Critical Care. Critical Care Delivery: The Importance of Process of Care and ICU Structure to Improved Outcomes: An Update From the American College of Critical Care Medicine Task Force on Models of Critical Care. Crit Care Med. 2015 Jul;43(7):1520-5. doi: 10.1097/CCM.0000000000000978. PMID 25803647
- [Derived] Sendagire C, Pisani L, Nuwagira A, Hewitt-Smith A, Nakibuuka J, Kiwalya H, Ayupo NC, Ogwal D, Kakaire D, Atumanya P, Khainza B, Nakayiza H, Nakandi H, Tomanya K, Alupo M, Ssemogerere L, Okello E, Lubikire A, Kintu A, Nyeko I, Kamau A, Kodippily C, Kwizera A, Beane A, Haniffa R, Salluh JIF. Potentially MOdifiable factors To ImproVe outcomes of mechanically Ventilated patients in a low-income country Intensive Care Units (MOTIVATE-ICU): rationale and protocol for a registry-embedded prospective observational study. Crit Care Sci. 2025 Oct 24;37:e20250273. doi: 10.62675/2965-2774.20250273. eCollection 2025. PMID 41259643